CLINICAL TRIAL: NCT01320774
Title: Efficacy, Tolerability and Handling of Daivobet® Gel in Patients With Psoriasis Vulgaris
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Collaborators: LEO Pharma GmbH, Neu-Isenburg, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: Treatment with Daivobet® Gel
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Daivobet® Gel — Once daily on areas with plaque psoriasis, treatment duration up to 8 weeks for body skin areas except scalp (scalp up to 4 weeks), treatment may be repeated under medical surveillance.

SUMMARY:
The purpose of this observational study is to evaluate the efficacy, tolerability, quality of life and handling of Daivobet® Gel by both physician and patient in daily practise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with light to moderate psoriasis vulgaris of trunk and extremities and treatment with Daivobet® Gel was planned anyway

Exclusion Criteria:

* Previous therapy with Daivobet® Gel
* Systemic therapy of psoriasis vulgaris
* Contraindications of Daivobet® Gel in the German package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting their attending dermatologist in the primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Handling of Daivobet® Gel | After appr 4 weeks
  Compared to previous topical treatment: Time required for application (previous treatment versus present treatment), time required until dressing is possible (previous treatment versus present treatment)

SECONDARY OUTCOMES:
Quality of life | 4 weeks
  Dermatology Life Quality Index (DLQI)
Physician's global Assessment of psoriasis vulgaris | 4 weeks
  6-step scale from "no visible disease (O)" to "very severe disease (5)
Side effects | 4 weeks
  number of participants with serious and non-serious adverse drug reactions, according to organ classes

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sticherling, Prof dr med, Principal Investigator — University clinic Erlangen-Nuernberg
Locations (1):
- University Clinic of Erlangen Nuernberg, Erlangen, Germany